CLINICAL TRIAL: NCT02507453
Title: Influence of Gravity on the Size-mass Illusion
Acronym: Massper
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-028
Record Dates: First submitted 2015-07-22; First posted 2015-07-24 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Influence of Gravity on the Size-mass Illusion (Other): to investigate the interaction between perceived size and perceived mass of objects in 0G and 1.8G compared to 1G using the size-mass illusion (SMI)
  Interventions: Other: parabolic flight; Other: mass/weight perception estimation; Device: ESA short-arm human centrifuge (SAHC)

INTERVENTIONS:
Other: parabolic flight
Other: mass/weight perception estimation — estimate the mass/weight perception, expressed by verbally report the absolute and relative mass of the object using a scale from 1 to 10 (1 being light and 10 being heavy)
Device: ESA short-arm human centrifuge (SAHC)

SUMMARY:
Parabolic flight is the only ground-based condition in which free-fall (0G) can be created long enough for safely testing changes in human perception and behavior. In addition to the 0G period, parabolic flight generates equal duration periods of 1.8G, which present another unique opportunity to test the same responses to hypergravity and back to 1G.

It is well known that performance decrements occur in astronauts during and after gravity level transitions. Illusions are commonly felt in orbit as well disorientation and perceptual limitations, mainly due to both psycho-physiological changes and adaptation and lack of familiar points of reference in the space environment. Studies performed during previous space missions showed several changes occurring in different gravity conditions, pointing out, for example, that colors and shadows were misleading, the depth and distance perception were weakened, and the linear perspective was lost. Visual perception is of primary importance for spatial orientation and object recognition because the static vestibular (otolithic) and proprioceptive signals are absent when free-floating. Consequently, astronauts become increasingly dependent on vision to perceive motion and orientation. All these factors play an important role in the adaptation of humans to spaceflight that needs to be analyzed to understand the underlying mechanisms that regulate human psycho-physiological adaptive process to changing gravity. Human psycho-physiological health has to be safeguarded and possibly improved when long-term human space missions are programmed in the near future.

The primary objective of this experiment is to investigate if the SWI illusion is present in altered gravity environments. Since weight cannot be estimated in 0G, investigators have developed a procedure during which the subject is asked to estimate the objects' mass by shaking them rather than lifting them. Our results in 1G indicate that a size-mass illusion (SMI) is also present in 1G. Our hypothesis is that the previously observed alteration in 3D visual perception in 0G, particularly in the height of 3D objects, as well as the change in proprioceptive inputs, will be responsible for changes in the SMI in 0G and 1.8G compared to 1G. In a separate proposal, investigators will also propose to perform this experiment using the ESA short-arm human centrifuge (SAHC), with subjects exposed to various centrifugal force levels, to further investigate the role of proprioceptive cues in the size-mass illusion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 21 to 65
* Right handed
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection.

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Pregnant women

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
perceived size and perceived mass of objects in 0G and 1.8G compared to 1G using the size-mass illusion (SMI) (composite) | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France